CLINICAL TRIAL: NCT01930539
Title: Treatment of Vitamin D Deficiency in Intestinal Rehabilitation Clinic Patients With a Portable Ultraviolet B Lamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0395-13-FB
Record Dates: First submitted 2013-08-14; First posted 2013-08-29 (Estimated); Results first posted 2023-08-25 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Vitamin D Deficiency; Short Bowel Syndrome
MeSH Terms: conditions — Vitamin D Deficiency; Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ultraviolet B lamp (Experimental): Intervention arm: Patients in the Ultraviolet B lamp group will continue vitamin D2/D3 daily and will receive 3 treatment sessions of Ultraviolet B light once a week for 12 weeks. Patients will receive Ultraviolet B light from Ultraviolet B lamp at a distance of 14 inches for duration of 5 minutes each area while wearing an Ultraviolet eye shield. Areas of skin exposure will include 3 different areas amounting to 27% of body surface area. 9% body surface area will include front of abdomen, lower back, each arm, each leg is 18%, each thigh. Ultraviolet B light sessions will be supervised and conducted by study personnel or Center for Clinical and Translational Research staff. A food questionnaire will be reviewed at each visit to assess dietary intake of calcium. Skin exam will be conducted at the beginning and end of the session.
  Interventions: Device: Ultraviolet B lamp
- Control (No Intervention): Patients in control group will continue with their current dose of Vitamin D2/D3 for 12 weeks.Patients will remain on the same steady dose for the duration of the study.These patients will not receive Ultraviolet B light sessions.

INTERVENTIONS:
Device: Ultraviolet B lamp — Ultraviolet-Fluorescent lamp (KBD, Inc, Crescent Springs, Kentucky, USA) was designed to use Ultraviolet B emitting fluorescent bulbs that have lower heat emission and allows a larger area of skin exposure. The Lamp is equipped with a timer for improved safety. This device is FDA (Food and Drug Administration) approved.
  Other Names: Sperti sunlamp "Del Sol"; Sperti, Crescent Springs, Kentucky
  Arms: Ultraviolet B lamp

SUMMARY:
This is a randomized, controlled, unblinded pilot study for patients with vitamin D deficiency in Intestinal Rehabilitation clinic. These patients are not able to absorb oral vitamin D efficiently and thus have a high prevalence of vitamin D deficiency, leading to low bone density.

The investigators will use FDA approved portable Ultraviolet B lamp for the intervention group, 11 patients will be recruited from October 2013 to end of January 2014 and study period is 12 weeks for each patient. Study completion will be end of April 2014.

Study hypothesis: Ultraviolet B light with a portable ultraviolet device will increase Total 25 hydroxy vitamin D level in Intestinal Rehabilitation Clinic patients.

DETAILED DESCRIPTION:
Vitamin D plays an integral role in bone metabolism and is one of the principal hormonal regulators of calcium and phosphorus absorption in the body. In 2011, the Endocrine Society defined Vitamin D deficiency as a 25 hydroxy vitamin D below 20 ng/ml and vitamin D insufficiency as a 25 hydroxy vitamin D of 21 ng/ml to 29 ng/ml.Without vitamin D, only 10 to 15% of dietary calcium and about 60% of phosphorus is absorbed.

Intestinal Rehabilitation clinic at University of Nebraska Medical Center includes patients with short bowel syndrome, multiple abdominal fistulae, and altered GI motility.

Hypovitaminosis D is associated with increased parathyroid hormone secretion,increased bone turnover, osteoporosis, histological osteomalacia and increased risk of hip and other fractures, and, in its most severe expression,clinical osteomalacia. These patients have been given high doses of both oral vitamin D2 and vitamin D3 supplementation without an improvement in vitamin D status due to poor intestinal absorption . Standardized treatment of vitamin D deficiency in most healthy individuals is achieved by giving vitamin D2 50,000 IU once a week for few weeks and then daily supplementation with lower doses. In the investigators Intestinal rehabilitation clinic, these patients are vitamin D insufficient or deficient while on large replacement doses of vitamin D2/D3 with some taking 200,000 IU daily.

It has been reported that irradiation with Ultraviolet B can be used safely and effectively to treat vitamin D deficiency among vitamin D deficient patients. Exposure of the body in a bathing suit to 1 Minimum Erythemal Dose (MED) of sunlight is equivalent to ingesting about 10,000 IU to 25,000 IU of vitamin D. Thus, exposure of 6% to 10% of the body surface to 1 MED is equivalent to ingesting about 600 to 2500 IU of vitamin D. Although ultraviolet irradiation can be achieved from exposure to sunlight, it is generally available only seasonally and difficult for persons who are too ill to spend much time outdoors. Ultraviolet-Fluorescent lamp (KBD, Inc, Crescent Springs, Kentucky,USA) was designed to use ultraviolet B emitting fluorescent bulbs that have lower heat emission and allows a larger area of skin exposure. The Lamp is equipped with a timer for improved safety. This device is FDA (Food and Drug Administration) approved.

Baseline labs include 25 hydroxy D, intact parathyroid hormone and complete metabolic profile. Patients will receive a 3 minute skin exposure to Ultraviolet B light and if they do not develop a sun burn, they will be randomized to Control or Ultraviolet B light group. Patients will continue their current dose of Vitamin D2/D3 for 12 weeks in both groups.Ultraviolet B light will be administered in 3 different areas on the same day for 5 minutes each, once a week at a distance of 14 inches wearing an UV eye shield. Areas of skin exposure will be based on rule of nine for body surface area which includes back, abdomen, thighs, and arms.

Patients will get blood draws at baseline and 12 weeks to monitor response to Ultraviolet B light. If Ultraviolet B light is able to increase total 25 hydroxy vitamin D level, it can potentially be used at home by these patients after receiving basic training and instructions.

ELIGIBILITY:
Inclusion Criteria:

* 25-hydroxy vitamin D level between 15ng/ml to 30mg/ml
* Age 19 years and above
* Patients on a stable dose of vitamin D2/D3 for last 3 months

Exclusion Criteria:

* Hypercalcemia (Serum Calcium (calculated) more than 1 mg/dl above the upper limit of normal i.e 11.3 mg/dl)
* Symptomatic Hypocalcemia (described as tetany )
* History of Sarcoidosis or Granulomatous diseases
* Patients on Calcitriol
* Liver failure defined as bilirubin more than 3, International Normalized Ratio of more than 3, Hepatic Transaminases 3 times of upper limit of normal, Decompensated cirrhosis with signs or icterus, varices, portal hypertension, encephalopathy.
* History of transplant or undergoing transplant evaluation
* Planned or Elective surgery in 6 months
* Personal or Family history of skin cancer
* History of photosensitivity
* Active skin disease in the areas planned for Ultraviolet B exposure
* Medications that limit sunlight exposure (such as tetracyclines or fluoroquinolones)
* Patients already undergoing tanning sessions
* Patients who are planning pregnancy or are breastfeeding
* Subjects with fair skin type I (Always burns easily, never tans)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn R Mack, MD, Principal Investigator — University of Nebraska Medical Center, Omaha
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Rosen CJ. Clinical practice. Vitamin D insufficiency. N Engl J Med. 2011 Jan 20;364(3):248-54. doi: 10.1056/NEJMcp1009570. No abstract available. PMID 21247315
- [Background] DiBaise JK, Young RJ, Vanderhoof JA. Intestinal rehabilitation and the short bowel syndrome: part 1. Am J Gastroenterol. 2004 Jul;99(7):1386-95. doi: 10.1111/j.1572-0241.2004.30345.x. PMID 15233682
- [Background] DiBaise JK, Young RJ, Vanderhoof JA. Intestinal rehabilitation and the short bowel syndrome: part 2. Am J Gastroenterol. 2004 Sep;99(9):1823-32. doi: 10.1111/j.1572-0241.2004.40836.x. PMID 15330926
- [Background] Armas LA, Dowell S, Akhter M, Duthuluru S, Huerter C, Hollis BW, Lund R, Heaney RP. Ultraviolet-B radiation increases serum 25-hydroxyvitamin D levels: the effect of UVB dose and skin color. J Am Acad Dermatol. 2007 Oct;57(4):588-93. doi: 10.1016/j.jaad.2007.03.004. Epub 2007 Jul 16. PMID 17637484
- [Background] Dabai NS, Pramyothin P, Holick MF. The effect of ultraviolet radiation from a novel portable fluorescent lamp on serum 25-hydroxyvitamin D3 levels in healthy adults with Fitzpatrick skin types II and III. Photodermatol Photoimmunol Photomed. 2012 Dec;28(6):307-11. doi: 10.1111/phpp.12000. PMID 23126292
- [Background] Chandra P, Wolfenden LL, Ziegler TR, Tian J, Luo M, Stecenko AA, Chen TC, Holick MF, Tangpricha V. Treatment of vitamin D deficiency with UV light in patients with malabsorption syndromes: a case series. Photodermatol Photoimmunol Photomed. 2007 Oct;23(5):179-85. doi: 10.1111/j.1600-0781.2007.00302.x. PMID 17803596
- [Background] Khazai NB, Judd SE, Jeng L, Wolfenden LL, Stecenko A, Ziegler TR, Tangpricha V. Treatment and prevention of vitamin D insufficiency in cystic fibrosis patients: comparative efficacy of ergocalciferol, cholecalciferol, and UV light. J Clin Endocrinol Metab. 2009 Jun;94(6):2037-43. doi: 10.1210/jc.2008-2012. Epub 2009 Mar 31. PMID 19336509
- See also: Portable Ultraviolet B lamp — http://www.sperti.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultraviolet B Lamp | Control
Started | 5 (participants) | 6 (participants)
Completed | 3 (participants) | 4 (participants)
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Adults age 19 and above with short bowel syndrome recruited from October 2013 to May 2014
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultraviolet B Lamp | Control | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 37 [30 to 58] | 50 [37 to 72] | 47 [30 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants] — Number of baseline participants
  participants
    United States | 3 | 4 | 7
Baseline vitamin D level [Mean (Standard Deviation); unit: ng/mL] — 25-hydroxy vitamin D level measured in ng/mL
  ng/mL | 19 (9) | 17 (7) | 18 (8)

OUTCOME MEASURES:

1. Primary Outcome: 25 Hydroxy Vitamin D Levels
Description: Our hypothesis is that Ultraviolet B light with a portable Ultraviolet device will increase Total 25 hydroxy vitamin D level in Intestinal Rehabilitation Clinic patients.
  We will measure serum level of 25 hydroxy vitamin D at baseline and 12 weeks to monitor the response of Ultraviolet B exposure administered by the portable Ultraviolet B lamp.
Time Frame: 12 weeks
Population: Male and female adults age 19 to 72
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Ultraviolet B Lamp | Control
Number analyzed (Participants) | 3 | 4
ng/mL
  Week 12 | 26 (14) | 14 (3)
  Week 0 | 19 (9) | 17 (7)

2. Secondary Outcome: Serum Intact Parathyroid Hormone Level
Description: Hypovitaminosis D is associated with increased Parathyroid hormone secretion (inversely related to 25 hydroxy D), increased bone turnover, osteoporosis, histological osteomalacia and increased risk of hip and other fractures, and, in its most severe expression,clinical osteomalacia.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Ultraviolet B Lamp | Control
Number analyzed (Participants) | 3 | 4
pg/ml
  Week 12 | 62 (59) | 70 (23)
  Week 0 | 139 (38) | 82 (30)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ultraviolet B Lamp | Control
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

LIMITATIONS AND CAVEATS:
The study population had variable bowel lengths impacting vitamin D absorption from oral supplements which were allowed but this did limit direct comparison of their vitamin D and parathyroid hormone (PTH) levels. Many had difficulty adhering to weekly visits leading to drop offs and small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No